CLINICAL TRIAL: NCT06601114
Title: The Effectiveness of Paracetamol Versus Ibuprofen in Management of Patent Ductus Arteriosus in Preterm Neonates
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arooj Khan (Other)
Responsible Party: Sponsor-Investigator, Arooj Khan, Head Of Paediatrics Sabir Khan, Khyber Teaching Hospital
Organization: Khyber Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 797/DME/KMC
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Patent Ductus Arteriosus in Preterm Infants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Paracetamol Group (Active Comparator): Group A: Paracetamol Group will receive Oral form of paracetamol with dosage of 15mg/kg every 6 hours for 3 days
  Interventions: Drug: Paracetamol Group
- Group B: Ibuprofen Group (Experimental): Group B: Ibuprofen Group will receive oral form of ibuprofen at initial dosage of 10mg/kg followed by 5mg/kg after 24 hours and 48 hours.
  Interventions: Drug: Ibuprofen group

INTERVENTIONS:
Drug: Paracetamol Group — Group A: Paracetamol Group will receive Oral form of paracetamol with dosage of 15mg/kg every 6 hours for 3 days
  Other Names: Experimental: Group B: Ibuprofen Group
  Arms: Group A: Paracetamol Group
Drug: Ibuprofen group — Group B: Ibuprofen Group will receive oral form of ibuprofen at initial dosage of 10mg/kg followed by 5mg/kg after 24 hours and 48 hours.
  Arms: Group B: Ibuprofen Group

SUMMARY:
This study aims to find and compare the effectiveness of paracetamol and ibuprofen in the closure of patent ductus arteriosus in preterm neonates.

The study is being conducted at Department of Nursery (special care baby unit) and Neonatal intensive care unit (NICU), KTH, Peshawar.

Neonates diagnosed with patent ductus arteriosus (PDA) in the Special care baby unit (SCBU) and Neonatal Intensive Care Unit (NICU) were enrolled in the study after obtaining ethical approval and informed consent from caretakers. The babies received routine care according to departmental policies. For PDA management, participants were randomly assigned to Group A, receiving oral paracetamol (Panadol, 15 mg/kg every 6 hours for 3 days), or Group B, receiving oral ibuprofen (Brufen, 10 mg/kg followed by 5 mg/kg after 24 and 48 hours). Paracetamol was defined as a selective COX-2 inhibitor, while ibuprofen was a non-selective COX inhibitor, both working by inhibiting prostaglandin synthesis. Procedures were supervised by a consultant pediatrician, with continuous patient monitoring. Treatment effectiveness, defined as complete PDA closure on echocardiography, was assessed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Neonates of gestational age more than 30 weeks and less than 37 weeks
* Neonates with birthweight of ≥1250g
* Neonates with postnatal age of 48-96 hours
* Neonates having one of the following echocardiographic criteria: a duct size > 2mm, a left atrium-to-aorta ratio >1.4, end diastolic reversal of blood flow in the aorta, or poor cardiac function in addition to clinical signs of patent ductus arteriosus

Exclusion Criteria:

* Gestational age less than 30 weeks and more than 37 weeks
* Presence of major congenital abnormalities
* Right-to-left ductal shunting
* Life-threatening infection
* Grade III or grade IV intraventricular hemorrhage
* Platelet count of <60000/mm3
* Hyperbilirubinemia requiring blood transfusion
* Persistent pulmonary hypertension

Ages: 48 Hours to 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 254 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Closure of Patent Ductus Arteriosus | 3 days
  The primary outcome is defined as the number of participants who achieve complete closure of the patent ductus arteriosus (PDA) after a course of the drug, as confirmed by echocardiography. Complete closure will be determined by the absence of ductal flow on color Doppler echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- MTI, Khyber Teaching Hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohlsson A, Shah PS. Paracetamol (acetaminophen) for patent ductus arteriosus in preterm or low-birth-weight infants. Cochrane Database Syst Rev. 2015 Mar 11;(3):CD010061. doi: 10.1002/14651858.CD010061.pub2. PMID 25758061
- [Background] Slaughter JL, Reagan PB, Newman TB, Klebanoff MA. Comparative Effectiveness of Nonsteroidal Anti-inflammatory Drug Treatment vs No Treatment for Patent Ductus Arteriosus in Preterm Infants. JAMA Pediatr. 2017 Mar 6;171(3):e164354. doi: 10.1001/jamapediatrics.2016.4354. Epub 2017 Mar 6. PMID 28046188
- [Background] Al-Lawama M, Alammori I, Abdelghani T, Badran E. Oral paracetamol versus oral ibuprofen for treatment of patent ductus arteriosus. J Int Med Res. 2018 Feb;46(2):811-818. doi: 10.1177/0300060517722698. Epub 2017 Sep 14. PMID 29239259
- [Derived] Shah SMA, Khan SA, Sadiq F, Gul R, Sadiq F, Khan MU, Khan MK, Uzma F, Khan A, Khan S. Comparison of the Effectiveness of Paracetamol and Ibuprofen in the Management of Patent Ductus Arteriosus in Preterm Neonates: A Randomized Controlled Trial. Mol Cell Pediatr. 2025 Jan 25;12(1):2. doi: 10.1186/s40348-025-00189-x. PMID 39862321